CLINICAL TRIAL: NCT03910894
Title: Health-related Quality of Life in Colon Cancer Patients
Brief Title: Health-related Quality of Life in Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Catarina Tiselius, Principal Investigator, Region Västmanland
Other Study IDs: HRQoL
Record Dates: First submitted 2019-03-31; First posted 2019-04-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-03

CONDITIONS: Health Related Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates health-related Quality of life in colon cancer patients in Västmanland, Sweden, at diagnosis, at 6 months, 1, 2 and 3 years after diagnosis, measured by the well-validated EORTC QLQ-C30 questionnaire.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

All patients diagnosed with colon cancer in Region Västmanland 2012-2016.

Exclusion Criteria:

Language problems, declined inclusion,

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with colon cancer in Region Västmanland 2012-2016, that accepted to be included in the study after written consent.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life | 2012-2016
  The EORTC QLQ-C30, a HRQoL questionnaire was used. It consists of 30 items comprising five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain). Six single items are also included (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties). The final two items in the questionnaire assess global health and overall QoL. Raw data were transformed to standardized scores ranging from 0 to 100 using the EORTC scoring manual. A high score on the functional scale represents a high level of functioning (i.e., higher is better), whereas a high score on the symptom scale represents a high level of symptoms (i.e., lower is better).

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Tiselius, PhD, Principal Investigator — Region Västmanland

IPD SHARING:
Plan to Share IPD: No
On request if suitable.

REFERENCES:
- [Derived] Tiselius C, Johansen F, Rosenblad A, Smedh K. Health-related quality of life is a significant prognostic factor for recurrence and overall survival in patients with colon cancer. BMC Cancer. 2025 Jun 10;25(1):1016. doi: 10.1186/s12885-025-14254-1. PMID 40495145
- [Derived] Tiselius C, Rosenblad A, Strand E, Smedh K. Risk factors for poor health-related quality of life in patients with colon cancer include stoma and smoking habits. Health Qual Life Outcomes. 2021 Sep 10;19(1):216. doi: 10.1186/s12955-021-01850-5. PMID 34507560